CLINICAL TRIAL: NCT04008836
Title: User Performance of the T-Plus Blood Glucose Monitoring Systems
Brief Title: User Performance of the Thunder Plus BGMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCA-PRO-2019-001-01
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; BGMS; blood glucose monitoring system; YSI Glucose Analyzer
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned to use the T-PLUS meter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Untrained Subjects WITH Diabetes use the T-PLUS BGMS (Experimental): Untrained subjects WITH Diabetes test capillary fingerstick and palm blood (and study staff test subject fingerstick blood) using the T-PLUS BGMS. All blood glucose results are compared to reference method results. Also, study staff test subject's venous blood and the blood glucose results are compared to the reference method results.
  Interventions: Device: T-PLUS Meter

INTERVENTIONS:
Device: T-PLUS Meter — Blood Glucose Monitoring System (BGMS)

SUMMARY:
T-PLUS (Thunder PLUS) is the code name of a blood glucose monitoring system (BGMS) consisting of a new meter and CONTOUR PLUS test strips. The meter can wirelessly transmit BG results using Bluetooth® Low Energy technology to the meter mobile application that will be available on specified versions of the iOS and Android mobile platforms.

This clinical trial will assess the performance (accuracy) of the T-PLUS meters by lay users enrolled as subjects in the study, and by health care professionals (also called study staff).

DETAILED DESCRIPTION:
This study is designed to satisfy both the FDA SMBG:2018 and the ISO 15197:2013, Section 8 requirements. Besides different analysis criteria, the main difference between these regulations is that FDA SMBG:2018 requires that both naïve users (people without diabetes) and people with diabetes to be included in the study population. The ISO 15197:2013 standard states that the study population shall only include people with diabetes.

The study will be conducted at one clinical site and enroll approximately 370 lay users. Ten to fifteen percent (10-15%) of the enrolled subjects will be people without diabetes and twenty percent (20%) of subjects enrolled with diabetes will have Type 1 diabetes.

Each subject will make one visit, lasting approximately 1 hour at the clinical site. Study sessions will be conducted by study staff members who have been trained on all aspects of the protocol.

PROCEDURES: Subjects will be assigned to use the T-PLUS meter and use one lot of Contour Plus test strip lots throughout the visit.

• Additional Procedures for Subjects with Diabetes: Subjects with diabetes will be given a venipuncture. The venous blood will be tested by the study staff using the T-PLUS system, and the YSI lab analyzer.

After all self-testing is completed, subjects with diabetes will be given a questionnaire to provide feedback about the new features of the system.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* Ability to speak, read and understand English. Subjects must demonstrate ability to read a paragraph from the first page of the UG to qualify for the study.
* Willing to complete all study procedures

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Pregnancy (self-reported)
* Physical, visual or neurological impairments that would make the person unable to perform testing with the BGMS.
* Previous participation in a blood glucose monitoring study using the Ascensia Contour TV3 or Thunder V3 and Thunder PLUS BGMS.
* Working for a medical laboratory, hospital or other clinical setting that involves training on or clinical use of blood glucose monitors.
* Being in this trial during or soon after xylose absorption testing (Xylose in the blood is known to cause interference). However, subjects can be enrolled as soon as 2 days after the test is performed (25 gms of oral xylose administered during this test is cleared within 480 mins or 8 hours).
* Working for a competitive medical device company, or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company.

  * Immediate family members are the subject's parents, spouse, children, and siblings, including the parent's spouse; step-children and adopted children and their spouses.
  * A competitive medical device company is a company that provides a medical device or components of a device that is related to diabetes.
* A condition, which in the opinion of the investigator or designee, would put the person or study conduct at risk. The reason for exclusion will be clearly documented by investigator or designee on the subject disposition form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research
Locations (1):
- Diablo Clinical Research (DCR), Walnut Creek, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from 10Jun2019 to 31Jul2019.
Period: Overall Study
Arm/Group | Untrained Subjects WITH Diabetes Use the T-PLUS BGMS
Started | 384
Completed | 384
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Subject Fingerstick Self Testing: Each subject performs fingerstick testing using the Thunder Plus meter.
Arm/Group | Subject Fingerstick Self Testing
Number analyzed (Participants) | 384
Age, Categorical [Count of Participants; unit: Participants] — count of number of subjects within an age range
  Participants
    <=18 years | 0
    Between 18 and 65 years | 269
    >=65 years | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (14.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224
  Male | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52
  Not Hispanic or Latino | 331
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 75
  White | 260
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 384

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Accurate BGMS Fingerstick Results
Description: Number of participants with results within ±15mg/dL of laboratory method at glucose concentration <100 mg/dL and within ±15% at glucose concentrations ≥100 mg/dL
Time Frame: One day
Measure: Count of Participants; unit: Participants
Arm/Group | Untrained Subjects WITH Diabetes Use the T-PLUS BGMS
Number analyzed (Participants) | 381
Participants | 373

2. Secondary Outcome: Number of Participants With Accurate BGMS Palm (AST) Results.
Description: Count of BGMS Palm (AST) from persons with diabetes within ±15mg/dL of laboratory method at glucose concentration <100 mg/dL and within ±15% at glucose concentrations ≥100 mg/d results
Time Frame: One day
Measure: Count of Participants; unit: Participants
Arm/Group | Untrained Subjects WITH Diabetes Use the T-PLUS BGMS
Number analyzed (Participants) | 365
Participants | 344

3. Secondary Outcome: Number of Responses to Questionnaire 1 That Are Within Specified Criteria.
Description: A Labeling evaluation (Ease of Use) was performed by the subjects who answered a survey to evaluate the ease of use of the test and the instructions in the package insert. A numerical score or rating will be reported by subjects for statement. The allowed response are 1) Strongly Disagree, 2) Disagree, 3) Neutral, 4) Agree, or 5) Strongly Agree. The number of responses for each statement that is 3,4, or 5 will be reported; 3,4, and 5 are considered favorable responses.
Time Frame: One day
Measure: Count of Participants; unit: Participants
Groups:
- Untrained Subjects WITH Diabetes Respond to a Questionnaire.: Untrained subjects WITH Diabetes respond to a questionnaire.
Arm/Group | Untrained Subjects WITH Diabetes Respond to a Questionnaire.
Number analyzed (Participants) | 332
Participants | 327

4. Secondary Outcome: Number of Participants With Accurate BGMS Venous Blood Results
Description: Number of participant's results from venous blood that are within 15% of the reference analyzer.
Time Frame: One day
Measure: Count of Participants; unit: Participants
Groups:
- Untrained Subjects WITH Diabetes Use the T-PLUS BGMS: Study staff test subject's venous blood and the blood glucose results are compared to the reference method results.
  T-PLUS Meter: Blood Glucose Monitoring System (BGMS)
Arm/Group | Untrained Subjects WITH Diabetes Use the T-PLUS BGMS
Number analyzed (Participants) | 327
Participants | 327

ADVERSE EVENTS:
Time Frame: Only collected on the day of the study
Description: No difference
Arm/Group | Untrained Subjects WITH Diabetes Use the T-PLUS BGMS
All-Cause Mortality (participants affected / at risk) | 0/384
Serious Adverse Events (participants affected / at risk) | 0/384
Other Adverse Events (participants affected / at risk) | 0/384

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study protocol and Statistical section (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT04008836/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT04008836/SAP_001.pdf